CLINICAL TRIAL: NCT01151839
Title: Preoperative Chemoradiation and Surgery Versus Surgery Alone in Squamous Cell Carcinoma of Oesophagus - A Randomized Controlled Trial
Brief Title: A Trial to Compare Preoperative Chemoradiation and Surgery Versus Surgery Alone in Squamous Cell Carcinoma of Oesophagus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Dr. Nikhil, AIIMS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IESC/T-186/2010
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-06

CONDITIONS: Esophageal Neoplasms
Keywords: Esophagus; squamous cell carcinoma; neoadjuvant chemoradiation
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Squamous Cell | interventions — Esophagectomy

ARMS (2):
- Surgery Alone (Active Comparator)
  Interventions: Procedure: Esophagectomy
- Neoadjuvant chemoradiation followed by surgery (Active Comparator)
  Interventions: Procedure: Neoadjuvant chemoradiation followed by surgery

INTERVENTIONS:
Procedure: Esophagectomy — Patient with squamous cell carcinoma of esophagus will be treated with surgery alone
  Arms: Surgery Alone
Procedure: Neoadjuvant chemoradiation followed by surgery — Patient with squamous cell carcinoma of esophagus will be treated by neoadjuvant chemoradiation followed by surgery
  Arms: Neoadjuvant chemoradiation followed by surgery

SUMMARY:
Carcinoma of the esophagus is the among the most common cancers in Indian population. While adenocarcinoma is more common in western countries, in India squamous cell carcinoma is the more frequent form. Surgery is the standard treatment in resectable lesions, but survival is poor. Adjuvant and neoadjuvant treatment therapy is used with an aim to improve the results. Though few randomized trials have addressed the issue of neoadjuvant chemoradiotherapy, the methodology was inhomogeneous and the populations studied were different. The investigators will be conducting a randomized controlled trial in patients with squamous cell carcinoma of the esophagus. Preoperative chemoradiation followed by surgery will be compared with surgery alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age < 65 years
2. Squamous cell carcinoma
3. Good performance status (Eastern Cooperative Oncology Group [ECOG] grades 0, 1 and 2)
4. Contrast enhanced computerized tomographic (CECT) scan suggesting a potentially resectable lesion. The features of resectability assessed on CECT scan will include - no evidence of infiltration of mediastinal structures such as the aorta (angle of contact <900, no obliteration of the triangular fat space between the esophagus, aorta, and spine), and pericardium20, and no evidence of tracheobronchial fistula or tumor extension into the airway lumen.
5. No evidence of distant metastasis on CECT.

Exclusion Criteria:

1. Patient refused consent for the study
2. Comorbid conditions which would preclude oesophagectomy

   * Poor performance status (ECOG > 2)
   * American Society of Anesthesiologists class IV
3. Metastatic disease detected on evaluation
4. Involvement of mediastinal structures except
5. Carcinoma involving cervical esophagus
6. Previous radiotherapy or chemotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Resectability rate | 2 years
  To compare the resectability rate of carcinoma esophagus between patients randomized to surgery alone and neoadjuvant chemoradiation followed by surgery
postoperative morbidity | 2 Years
  To compare the postoperative morbidity between patients of carcinoma esophagus randomized to surgery alone versus chemoradiation followed by surgery
operative mortality | 2 Years
  To compare the operative mortality between patients randomized to surgery alone and neoadjuvant chemoradiation followed by surgery.

SECONDARY OUTCOMES:
Early disease control | 2 years
  To compare the early disease control in patients randomized to receive either neoadjuvant chemoradiation and surgery or surgery alone.
Treatment toxicity | 2 years
  This study will also assess the treatment toxicity of preoperative chemoradiation

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil -, MS, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India